CLINICAL TRIAL: NCT02525562
Title: Stryker NTX Registry Scorpio NRG Triathlon Total Knee, Triathlon PKR With X3 Insert International Multicentre Outcomes Register
Brief Title: Stryker NTX Registry Scorpio NRG (Re-"Energize"), Triathlon Total Knee, Triathlon Partial Knee Resurfacing (PKR) With X3 Polyethylene Insert
Acronym: NTX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-S-044
Record Dates: First submitted 2015-06-11; First posted 2015-08-17 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Scorpio NRG Total Knee System (Other): Patients eligible for Scorpio NRG Total Knee System with X3 insert
  Interventions: Device: Scorpio NRG Total Knee System with X3 insert; Procedure: Total Knee Replacement
- Triathlon Total Knee System (Other): Patients eligible for Triathlon Total Knee System with X3 insert
  Interventions: Device: Triathlon Total Knee System with X3 insert; Procedure: Total Knee Replacement
- Triathlon Partial Knee Resurfacing (Other): Patients eligible for Triathlon PKR System with X3 insert
  Interventions: Device: Triathlon PKR System with X3 insert; Procedure: Partial Knee Resurfacing

INTERVENTIONS:
Device: Triathlon Total Knee System with X3 insert — Total knee replacement
  Arms: Triathlon Total Knee System
Device: Scorpio NRG Total Knee System with X3 insert — Total knee replacement
  Arms: Scorpio NRG Total Knee System
Device: Triathlon PKR System with X3 insert — Partial Knee Resurfacing
  Arms: Triathlon Partial Knee Resurfacing
Procedure: Total Knee Replacement — Total Knee Replacement
  Arms: Scorpio NRG Total Knee System; Triathlon Total Knee System
Procedure: Partial Knee Resurfacing — Partial Knee Resurfacing
  Arms: Triathlon Partial Knee Resurfacing

SUMMARY:
Provide outcomes information with regard to surgical and implant performance and patient clinical outcomes of the patients who are eligible for either a Total Knee Arthroplasty (TKA) replacement surgery or Partial Knee Resurfacing (unicompartmental knee arthroplasty, UKA)

DETAILED DESCRIPTION:
The objective of this registry is to provide outcomes information with regard to surgical and implant performance and patient clinical outcomes of the patients who are eligible for a either a Total Knee Arthroplasty (TKA) replacement surgery involving the Scorpio NRG or Triathlon Total Knee System or Triathlon PKR Partial Knee Resurfacing (unicompartmental knee arthroplasty, UKA), all of which with X3 inlay. The register will follow the standard clinical procedures used by the institutions for patient selection for knee arthroplasty surgery, patient surgery and patient follow-up. Therefore there will be, with regard to this register, no additional assessment, examination, procedure or follow-up visits compared to those usually performed in the institution (routine standard normal procedures).

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring primary TKA, suitable for the use of the Scorpio NRG with X3 insert or Triathlon Total Knee System with X3 insert, or, patients requiring partial knee resurfacing (unicompartmental knee) suitable for the use of the Triathlon PKR (Partial Knee Resurfacing) System with X3 insert
2. Patients who understand the conditions of the outcomes registry and are willing and able to comply with the standard post-operative evaluations and the prescribed rehabilitation.
3. Patients who signed the Informed Consent Form (approved by Ethics Committee if required) prior to surgery.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2012-06-28 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Romain Seil, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (3):
- Kliniken Dr. Erler gGmbH, Nuremberg, Bavaria, Germany
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Worcestersire Acute Hospital NHS Trust, Alexandra Hospital, Redditch, Worcestersire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 237 participants enrolled - 14 participants censored = 223 participants followed. All participants received a Triathlon Total Knee Replacement. No participants received a Scorpio NRG Total Knee Replacement or a Triathlon Partial Knee Resurfacing Replacement.
Period: Overall Study
Arm/Group | Triathlon Total Knee System | Scorpio NRG Total Knee System | Triathlon Partial Knee Resurfacing
Started | 223 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 223 | 0 | 0
Not completed — Death | 9 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0
Not completed — Withdrawal by Subject | 37 | 0 | 0
Not completed — Revision/Removal of Study Device | 4 | 0 | 0
Not completed — Study Closed by Sponsor | 154 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes participants who received the Triathlon Total Knee System and were not censored from analysis.
Arm/Group | Triathlon Total Knee System
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.61 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Luxembourg | 30
  United Kingdom | 100
  Germany | 93

OUTCOME MEASURES:

1. Primary Outcome: Survivorship of the Device
Description: Survivorship shown in Kaplan Meier survival curves (statistic used to estimate the survival function from lifetime data).
Time Frame: Preoperative to 1 year, 1 year, 3 years, and 5 years. Survivorship is unavailable at 10 years due to study termination.
Population: This primary outcome measure (10 year) was not analyzed due to termination of the study. Results display number of participants at each timepoint (i.e., preoperative to 1 year, 1 year, 3 years, and 5 years) that remain free from revision; 10 year not reported due to study termination. Overall number of participants analyzed is based upon the preoperative to 1 year population, originally 223 participants with 4 early terms (no surgery), therefore n=219.
Measure: Number; unit: participants free from revision
Arm/Group | Triathlon Total Knee System
Number analyzed (Participants) | 219
participants free from revision
  Free from Revision at Preoperative to 1 year | 218
  Free from Revision at 1 year: number analyzed (Participants) | 211
  Free from Revision at 1 year | 207
  Free from Revision at 3 years: number analyzed (Participants) | 175
  Free from Revision at 3 years | 170
  Free from Revision at 5 years: number analyzed (Participants) | 155
  Free from Revision at 5 years | 150

2. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Society Score (KSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability (Pain/Motion KSS subscale is 0 to 100, with 100 representing a better outcome), and one for functional parameters (Function KSS subscale is 0 to 100, with 100 representing a better outcome). Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points, and Combined KSS is the summed average of the Pain/Motion and Function sub-scores, leading to a Combined KSS total ranging from 0 to 200 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: Pre-operative, 1, 3, and 5 years. The KSS for 7 and 10 year timepoints are unavailable due to study termination.
Population: Participants with available data through 5 years. Overall number of participants analyzed is based upon the pre-operative population that completed a KSS evaluation. One participant did not have data KSS data available at the preoperative timepoint (n=222).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon Total Knee System
Number analyzed (Participants) | 222
units on a scale
  Combined KSS Mean Preoperative Score (0-200 points) | 101.1 (26.53)
  Combined KSS Mean 1 Year Score (0-200 points): number analyzed (Participants) | 212
  Combined KSS Mean 1 Year Score (0-200 points) | 155.32 (29.82)
  Combined KSS Mean 3 Year Score (0-200 points): number analyzed (Participants) | 168
  Combined KSS Mean 3 Year Score (0-200 points) | 161.4 (30.03)
  Combined KSS Mean 5 Year Score (0-200 points): number analyzed (Participants) | 150
  Combined KSS Mean 5 Year Score (0-200 points) | 158.03 (29.32)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Injury and Osteoarthritis Outcome Score (KOOS) Patient Questionnaire.
Description: KOOS consists of 5 subscales: Symptoms, Pain, Function in Daily Living, Function in Sport and Recreation, and knee related Quality of Life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given for each subscale (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score is calculated for each subscale, with a minimum of 0 indicating extreme symptoms and a maximum of 100 indicating no symptoms. Only subscale scores are reported.
Time Frame: Pre-operative, 1, 3, and 5 years. The KOOS for 7 and 10 year timepoints are unavailable due to study termination.
Population: Participants with available data through 5 years. Overall number of participants analyzed is based upon the pre-operative population. The Function in Sport and Recreation, Number of Analyzed Participants at 3-years and 5-years is lower than other subscales due to participants not selecting a box on the Likert scale at these timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon Total Knee System
Number analyzed (Participants) | 223
units on a scale
  Symptoms: KOOS Mean Preoperative Score | 45.95 (19.96)
  Symptoms: KOOS Mean 1 Year Score: number analyzed (Participants) | 210
  Symptoms: KOOS Mean 1 Year Score | 78.96 (16.42)
  Symptoms: KOOS Mean 3 Year Score: number analyzed (Participants) | 173
  Symptoms: KOOS Mean 3 Year Score | 81.05 (17.23)
  Symptoms: KOOS Mean 5 Year Score: number analyzed (Participants) | 151
  Symptoms: KOOS Mean 5 Year Score | 81.43 (16.7)
  Pain: KOOS Mean Preoperative Score | 40.02 (17.51)
  Pain: KOOS Mean 1 Year Score: number analyzed (Participants) | 210
  Pain: KOOS Mean 1 Year Score | 81.2 (17.59)
  Pain: KOOS Mean 3 Year Score: number analyzed (Participants) | 173
  Pain: KOOS Mean 3 Year Score | 82.28 (19.93)
  Pain: KOOS Mean 5 Year Score: number analyzed (Participants) | 151
  Pain: KOOS Mean 5 Year Score | 82.02 (19.98)
  Function, Daily Living: KOOS Mean Preoperative Score | 43.05 (19.27)
  Function, Daily Living: KOOS Mean 1 Year Score: number analyzed (Participants) | 210
  Function, Daily Living: KOOS Mean 1 Year Score | 79.28 (18.68)
  Function, Daily Living: KOOS Mean 3 Year Score: number analyzed (Participants) | 173
  Function, Daily Living: KOOS Mean 3 Year Score | 80.33 (20.68)
  Function, Daily Living: KOOS Mean 5 Year Score: number analyzed (Participants) | 151
  Function, Daily Living: KOOS Mean 5 Year Score | 78.86 (21.38)
  Function, Sports and Recreational: KOOS Mean Preoperative Score | 14.46 (19.93)
  Function, Sports and Recreational: KOOS Mean 1 Year Score: number analyzed (Participants) | 210
  Function, Sports and Recreational: KOOS Mean 1 Year Score | 47.24 (29.27)
  Function, Sports and Recreational: KOOS Mean 3 Year Score: number analyzed (Participants) | 172
  Function, Sports and Recreational: KOOS Mean 3 Year Score | 52.11 (30.86)
  Function, Sports and Recreational: KOOS Mean 5 Year Score: number analyzed (Participants) | 148
  Function, Sports and Recreational: KOOS Mean 5 Year Score | 50.42 (30.65)
  Quality of Life: KOOS Mean Preoperative Score | 23.12 (17.22)
  Quality of Life: KOOS Mean 1 Year Score: number analyzed (Participants) | 210
  Quality of Life: KOOS Mean 1 Year Score | 67.11 (25.33)
  Quality of Life: KOOS Mean 3 Year Score: number analyzed (Participants) | 173
  Quality of Life: KOOS Mean 3 Year Score | 67.02 (27.19)
  Quality of Life: KOOS Mean 5 Year Score: number analyzed (Participants) | 151
  Quality of Life: KOOS Mean 5 Year Score | 69.77 (26.17)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the EuroQuol-5 Dimension Health Questionnaire (EQ-5D) Patient Questionnaire.
Description: The EuroQol-5 Dimension (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; EQ-5D descriptive system and the visual analogue scale (VAS).
  The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
  With the EQ VAS, the respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: Pre-operative, 1, 3, and 5 years. The EQ-5D for 7 and 10 year timepoints is unavailable due to study termination.
Population: Participants with available data through 5 years. Overall number of participants analyzed is based upon the pre-operative population with EQ-5D data available. Number of Analyzed Participants at the Preoperative timepoint for this assessment (EQ-5D) is fewer than overall due to two participants not completing the preoperative questionnaire, therefore n=221.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon Total Knee System
Number analyzed (Participants) | 221
units on a scale
  Descriptive EQ-5D: Mean Preoperative Score | 0.42 (0.33)
  Descriptive EQ-5D: Mean 1 Year Score: number analyzed (Participants) | 210
  Descriptive EQ-5D: Mean 1 Year Score | 0.76 (0.26)
  Descriptive EQ-5D: Mean 3 Year Score: number analyzed (Participants) | 173
  Descriptive EQ-5D: Mean 3 Year Score | 0.77 (0.26)
  Descriptive EQ-5D: Mean 5 Year Score: number analyzed (Participants) | 151
  Descriptive EQ-5D: Mean 5 Year Score | 0.76 (0.27)
  EQ-5D VAS: Mean Preoperative Score | 62 (21.9)
  EQ-5D VAS: Mean 1 Year Score: number analyzed (Participants) | 210
  EQ-5D VAS: Mean 1 Year Score | 74.7 (19.1)
  EQ-5D VAS: Mean 3 Year Score: number analyzed (Participants) | 173
  EQ-5D VAS: Mean 3 Year Score | 73.6 (19.8)
  EQ-5D VAS: Mean 5 Year Score: number analyzed (Participants) | 151
  EQ-5D VAS: Mean 5 Year Score | 71.5 (19.5)

ADVERSE EVENTS:
Time Frame: All operative site and general medical adverse events, as well as elective surgery involving other joints, over the course of the 5-year surveillance period (original 10 years surveillance, however, study terminated early).
Description: Censored were not included as at risk. Date of occurrence, date diagnosed, type of complication and treatment were collected. Industry standard Adverse Event (AE) and Serious Adverse Event) SAE terms were used in this study.
Groups:
- Operative Adverse Events; Non-operative Adverse Events: Triathlon Total Knee System with X3 insert, reported by participant.
Arm/Group | Operative Adverse Events | Non-operative Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/223 | 9/223
Serious Adverse Events (participants affected / at risk) | 18/223 | 55/223
Other Adverse Events (participants affected / at risk) | 0/223 | 52/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=223) | Non-operative Adverse Events (N=223)
Non-operative (Cardiac disorders) | 0/0 (0) | 11 (11)
Non-Operative (Eye disorders) | 0/0 (0) | 1 (1)
Non-Operative (Gastrointestinal disorders) | 0/0 (0) | 6 (6)
Operative (Infections and infestations) | 1 (1) | 0/0 (0)
Non-Operative (Infections and infestations) | 0/0 (0) | 1 (1)
Operative (Injury, poisoning and procedural complications) | 2 (2) | 0/0 (0)
Operative (Musculoskeletal and connective tissue disorders) | 13 (13) | 0/0 (0)
Non-Operative (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 16 (18)
Non-Operative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 9 (9)
Non-Operative (Nervous system disorders) | 0/0 (0) | 1 (1)
Non-Operative (Renal and urinary disorders) | 0/0 (0) | 4 (5)
Non-Operative (Reproductive system and breast disorders) | 0/0 (0) | 1 (1)
Operative (Skin and subcutaneous tissue disorders) | 2 (2) | 0/0 (0)
Non-Operative (Vascular disorders) | 0/0 (0) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=223) | Non-operative Adverse Events (N=223)
Elective Procedures (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 41 (47)
Non-Operative (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 11 (11)

LIMITATIONS AND CAVEATS:
The study was terminated at the 5-year timepoint, therefore the primary outcome measure of survivorship of the device at 10-years was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Principal Investigators and the Sponsor (or its agents) that requires Investigators to allow Sponsor at least 30 days to review material intended for publications in order to redact any Confidential Information or Inventions therefrom.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02525562/Prot_SAP_000.pdf